CLINICAL TRIAL: NCT05869877
Title: The PIV5Rights Safety and Quality Bundle
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Vygon GmbH & Co. KG (Industry)
Responsible Party: Principal Investigator, Lee Steere, Nurse Manager IV Therapy Services, Hartford Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: HHC-2022-0276
Record Dates: First submitted 2023-05-09; First posted 2023-05-22 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Catheter Complications

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial evaluating a peripheral intravenous catheter (PIVC) inserting using a bundled approach. Will evaluate the for extended dwell time and less complications compared to a PIVC using a non-bundled approach
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (No Intervention): Proficient RN who works in IV Therapy Department - PIVC inserted without using ultrasound; non-bordered transparent dressing; 1-1.25 inch catheter; microbore extension set with neutral needleless connector; transpore tape. Standard of care
- Bundled (Experimental): Proficient RN who works in IV Therapy Department - 6 cm catheter inserted with or without ultrasound; chlorhexidine embedded transparent bordered dressing; transpore tape; microbore extension set with antireflux needleless connector
  Interventions: Device: Bundled

INTERVENTIONS:
Device: Bundled — An peripheral intravenous catheter will be inserted by an RN specially trained in PIVC placement, with or without ultrasound. Using best of class medical products, will evaluate dwell time and complications of the PIVC inserted using a bundled approach versus one inserted with the bundle
  Arms: Bundled

SUMMARY:
Purpose of this study is to see if a Peripheral Intravenous Catheter PIVC will last longer if inserted by a Registered Nurse (RN) who specializes in inserting PIVCs. Main question it aims to answer:

1. We believe that the use of the ultrasound, an RN who specializes in PIVC placement with the use of ultrasound and the use of best of class medical technology, may improve first stick success with PIVC insertion and the length of time the PIVC stays in place without showing any related complications

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent, patients will be randomized using Research Randomizer. At that time, the IV Therapist will insert a PIVC using standard of care medical equipment (control) or use ultrasound guidance, if needed, to insert a PIVC using the bundle with the best of class medical devices. Daily, a research RN will round, assess the site and take a picture. When therapy is complete or the PIVC malfunctions, the research RN will document the reason why the PIVC failed and that patient will no longer remain in the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older with not upper limit
* requires an IV for fluid and or medication administration
* able to read and write English and willing to complete written, informed consent

Exclusion Criteria:

* Unable to speak and read English
* Vulnerable populations such as minors (under age of 18)
* Incompetent or mentally challenged
* Prisoners
* Pregnant women or the unborn
* presented in the hospital prior to study start date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-03-25 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
1 PIVC Per Patient Stay | 1 year
  To compare the proportion of patients for whom the initial catheter insertion is sufficient for their duration of care across the two groups

SECONDARY OUTCOMES:
Dwell Time | 1 year
  To compare dwell times between the 2 groups. Dwell time is defined as the time from line insertion to line removal.
Cost Impact | 1 year
  To compare cost with additional PIVC's inserted if PIVC failed to make it until the end of therapy
Outcome Analysis | 1 year
  To compare IV related complications between the 2 groups (infiltrations, occlusions, phlebitis)

CONTACTS AND LOCATIONS:
Overall Officials: Lee J Steere, ADN, Principal Investigator — Hartford Hospital